CLINICAL TRIAL: NCT03327389
Title: Effect of Dexmedetomidine on Renal Function and Delayed Graft Function After Kidney Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2017-0767
Record Dates: First submitted 2017-10-23; First posted 2017-10-31 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: 1. Dexmedetomidine group
  2. Control group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: participants, investicator, outcome assessors will be blinded for group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Group D) (Experimental): Dexmedetomidine infusion during surgery Dexmedetomidine was infused at a rate of 0.4 μg/kg/h starting immediately after anesthetic induction and continued until skin closure
  Interventions: Drug: Dexmedetomidine
- Control (Group C) (Placebo Comparator): 0.9% NaCl infusion during surgery 0.9% NaCl was infused at a rate of 0.4 μg/kg/h starting immediately after anesthetic induction and continued until skin closure
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine was infused at a rate of 0.4 μg/kg/h starting immediately after anesthetic induction and continued until skin closure.
  Arms: Dexmedetomidine (Group D)
Drug: placebo — 0.9% NaCl was infused at a rate of 0.4 μg/kg/h starting immediately after anesthetic induction and continued until skin closure
  Arms: Control (Group C)

SUMMARY:
The purpose of this study is to elucidate the effect of dexmedetomidine on renal function and delayed graft function after kidney transplantation

ELIGIBILITY:
Inclusion Criteria:

1. adult (20-80 years old)
2. patients undergoing elective kidney transplantation

Exclusion Criteria:

1. emergency surgery
2. severe sinus bradycardia (<50 beats per min [bpm])
3. second-degree or third-degree heart block
4. decreased heart function (EF <30%)
5. acute myocardial ischemia
6. serious hepatic dysfunction (Child-Pugh class C)
7. patients with known or suspected severe adverse reactions to DEX (or clonidine)
8. treatment with clonidine or dexmedetomidine in the past 30 days

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-09-28 (Estimated); Study Completion 2019-09-28 (Estimated)

PRIMARY OUTCOMES:
Serum creatinine level | postoperative 7 day

SECONDARY OUTCOMES:
incidence of delayed graft function | 7 days after surgery
level of serum creatinine | maximum 30 days before surgery, 1 hour after surgery, 1 day, 2 day, 3 day, 5 day, 7 day after surgery
blood urea nitrogen (BUN) | maximum 30 days before surgery, 1 hour after surgery, 1 day, 2 day, 3 day, 5 day, 7 day after surgery
cystatin C | maximum 30 days before surgery, 1 hour after surgery, 1 day, 2 day, 3 day, 5 day, 7 day after surgery
Neutrophil gelatinase-associated lipocalin (NGAL) | maximum 30 days before surgery, 1 hour after surgery, 1 day, 2 day, 3 day, 5 day, 7 day after surgery
urine output | during surgery, 1 day, 2 day, 3 day, 4 day, 5 day, 6 day, 7 day after surgery
fluid intake(intraoperative intake and output measured by the amount of fluid(crystalloid/colloid)(mL) and blood administered(mL)) | during surgery, 1 day, 2 day, 3 day, 4 day, 5 day, 6 day, 7 day after surgery
kidney ultrasound | 1 week, 1 month after surgery, if possible
inflammatory mediator (IL-18, Il-1b) level | immediately after induction, immediately after vessel clamp, immediately after reperfusion, 1hour after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park JH, Koo BN, Kim MS, Shin D, Kwak YL. Effects of intraoperative dexmedetomidine infusion on renal function in elective living donor kidney transplantation: a randomized controlled trial. Can J Anaesth. 2022 Apr;69(4):448-459. doi: 10.1007/s12630-021-02173-1. Epub 2021 Dec 20. PMID 34931289